CLINICAL TRIAL: NCT05551052
Title: Prospective, Multi-center Observational Study for the Clinical Validation of the Next Generation Test for Blood-based Screening of Colorectal Cancer
Brief Title: CRC Detection Reliable Assessment With Blood
Acronym: CRC-DRAW
Status: Active, not recruiting | Type: Observational
Sponsor: New Day Diagnostics (Network)
Responsible Party: Sponsor
Other Study IDs: SPR0033P
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Adenomas Colon; Colon Cancer; Rectal Cancer; Colon Neoplasm; Colon Lesion; Colon Disease; Colon Polyp; Polyps; Adenoma; Rectal Diseases; Rectal Polyp; Gastrointestinal Neoplasms; Intestinal Neoplasms; Colonic Diseases, Functional; Intestinal Disease
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Colonic Diseases; Colonic Polyps; Polyps; Adenoma; Rectal Diseases; Gastrointestinal Neoplasms; Intestinal Neoplasms; Colonic Diseases, Functional; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be de-identified and used to validate the performance characteristics of the Next-Gen CRC Screening Test. Blood samples may also be used for future research and development, feasibility and validation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Next-Gen CRC Screening Test: Adults 45 years of age and older who are at average risk of developing colorectal cancer and eligible for a screening colonoscopy
  Interventions: Diagnostic Test: Next-Gen CRC Screening Test

INTERVENTIONS:
Diagnostic Test: Next-Gen CRC Screening Test — The Next-Gen CRC Screening Test is a blood-based screening test for detection of CRC.

SUMMARY:
The CRC DRAW study will assess the sensitivity and specificity of the blood-based, Next-Gen CRC Screening Test for the detection of CRC.

DETAILED DESCRIPTION:
The CRC DRAW study is a prospective, multi-center, observational study to validate the Next-Gen CRC Screening test for the detection of CRC. The study will collect blood samples from average-risk participants scheduled for screening colonoscopies.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 45 years of age or older at time of enrollment.
2. Participant is at average risk for development of colorectal cancer (as defined by inclusion and exclusion criteria)
3. Participant is able and willing to undergo a screening colonoscopy
4. Participant is able and willing to sign informed consent and adhere to study requirements
5. Participant is able to provide blood sample prior to colonoscopy (within 90 days of scheduled colonoscopy).

Exclusion Criteria:

1. Previous personal history of CRC or precancerous lesions
2. Positive result from non-invasive screening test within the associated recommended intervals:

   2.1 Fecal occult blood test or fecal immunochemical test within the previous 12 months 2.2 Epi proColon test within the previous 12 months 2.3 FIT-DNA (Cologuard) test within the previous 36 months
3. Diagnosed with condition associated with higher risk for colorectal cancer, such as:

   3.1 Inflammatory bowel disease (IBD) 3.2 Chronic ulcerative colitis (CUC) 3.3 Crohn's disease 3.4 Familial adenomatous polyposis (FAP) 3.5 Familial history for colorectal cancer 3.5.1 One or more first-degree relatives diagnosed with CRC or adenomatous polyps before 60 years of age 3.5.2 Two or more first degree relatives diagnosed at any age with CRC
4. Individuals with relevant familial (hereditary) cancer syndrome, such as:

   4.1 Hereditary non-polyposis colorectal cancer syndrome (HNPCC or Lynch Syndrome) 4.2 Peutz-Jeghers Syndrome 4.3 MYH-Associated Polyposis (MAP) 4.4 Gardner's syndrome 4.5Turcot's (or Crail's) syndrome 4.6 Cowden's syndrome, 4.7Juvenile Polyposis 4.8 Cronkhite-Canada syndrome 4.9 Neurofibromatosis 4.10 Familial Hyperplastic Polyposis
5. Diagnosed with chronic gastritis or cirrhosis
6. Current diagnosis of any cancer, except non-melanoma skin cancer
7. Overt rectal bleeding or bleeding hemorrhoids within previous 30 days
8. A colonoscopy within the previous 9 years, with the exception of a failed colonoscopy due to poor bowel preparation
9. Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 45 years of age and older who are at average risk of developing colorectal cancer and eligible for a screening colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for CRC of the Next-Gen CRC Screening Test | blood collection up to 90 days from colonoscopy
  Clinical Performance
Specificity for CRC of the Next-Gen CRC Screening Test | blood collection up to 90 days from colonoscopy
  Clinical Performance

SECONDARY OUTCOMES:
Sensitivity for advanced precancerous lesions of the Next-Gen CRC Screening Test | blood collection up to 90 days from colonoscopy
  Clinical Performance
Specificity for no colorectal neoplastic findings of the Next-Gen CRC Screening Test | blood collection up to 90 days from colonoscopy
  Clinical Performance

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Gastro SB, Chula Vista, California
  - SDG Clinical Research, San Diego, California
  - Medical Associates Research Group, San Diego, California

IPD SHARING:
Plan to Share IPD: No